CLINICAL TRIAL: NCT02899936
Title: Community Based Safety Study of 2-drug (Diethylcarbamazine and Albendazole) Versus 3-drug (Ivermectin, Diethylcarbamazine and Albendazole) Therapy for Lymphatic Filariasis
Brief Title: Death to Onchocerciasis and Lymphatic Filariasis (DOLF) Triple Drug Therapy for Lymphatic Filariasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Case Western Reserve University (Other); Indian Council of Medical Research (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201607068
Record Dates: First submitted 2016-08-22; First posted 2016-09-14 (Estimated); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Lymphatic Filariasis
Keywords: Mass drug administration; Safety Data
MeSH Terms: conditions — Elephantiasis, Filarial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 drug dose - DA (Active Comparator): Drug treatment with two-drug regimen diethylcarbamazine and albendazole (DA)
  Interventions: Drug: 2 drug dose - DA
- 3 drug dose - IDA (Experimental): Triple-drug regimen Ivermectin, diethylcarbamazine and albendazole (IDA)
  Interventions: Drug: 3 drug dose - IDA

INTERVENTIONS:
Drug: 3 drug dose - IDA — Lymphatic Filariasis Mass Drug Administration (MDA) with triple drug therapy of ivermectin, diethylcarbamazine, and albendazole (IDA)
  Other Names: IDA
  Arms: 3 drug dose - IDA
Drug: 2 drug dose - DA — Lymphatic Filariasis Mass Drug Administration (MDA) with the currently used standard of care combination drug therapy of diethylcarbamazine, and albendazole (DA)
  Other Names: DA
  Arms: 2 drug dose - DA

SUMMARY:
The DOLF Triple Drug Therapy for Lymphatic Filariasis study will determine the frequency, type and severity of adverse events following triple-drug therapy (IVM+DEC+ALB, IDA) compared to the standard two-drug treatment (DEC+ALB, DA) in infected and uninfected individuals in a community in 5 different countries. The objective is to acquire safety, efficacy, and acceptability data to assess the safety and acceptability of the IDA drug combination.

DETAILED DESCRIPTION:
In 2000, the World Health Organization (WHO) launched the Global Programme to Eliminate Lymphatic Filariasis (GPELF) to eliminate lymphatic filariasis as a public health problem by 2020. To interrupt transmission, WHO recommends therapy using combinations of two medicines delivered to entire at-risk populations through a strategy known as mass drug administration. Ivermectin (IVM) and albendazole (ALB) are administered in areas where onchocerciasis is co-endemic; diethylcarbamazine (DEC) and albendazole (ALB) are administered in areas where onchocerciasis is not co-endemic.

Results of a pilot study in Papua New Guinea suggest that triple drug therapy (ivermectin, diethylcarbamazine and albendazole) is superior to the currently recommended two-drug regimen (DEC+ALB, DA). A single dose of the triple therapy (IVM+DEC+ALB, IDA) rapidly achieved complete clearance of Wuchereria bancrofti microfilariae from the blood of 12 individuals for at least one year post-treatment. All six individuals tested at 24 months were still amicrofilaremic, suggesting that the triple therapy might permanently sterilizes adult filarial worms. Many people treated in these studies experienced transient systemic adverse events commonly associated with diethylcarbamazine or ivermectin treatment of filariasis. Adverse events were more frequent after the triple therapy than after the usual combination of two drugs. However, no serious adverse events were observed. The dramatic reduction and sustained decrease of microfilaria along with the safety profile seen in the Papua New Guinea studies suggest that the triple drug therapy may be a useful tool to achieve the goal of eliminating lymphatic filariasis as a public health problem by 2020.

Although the study cited above has clearly demonstrated the superiority of the triple therapy for clearing W. bancrofti microfilaria from the blood, more safety and efficacy data are needed before triple therapy can be rolled out on a large scale as a mass drug administration regimen in lymphatic filariasis endemic countries. WHO recommends a best practice called "cohort event monitoring" for demonstrating safety of new drug regimens for public health program use. Establishing safety through such methodology requires pre and post treatment assessment from at least 10,000 people treated with the triple therapy across multiple settings.

It is therefore proposed to conduct a cohort event monitoring study to acquire safety data. Efficacy and acceptability components will also be included in the study. Similar studies will be conducted simultaneously in Haiti, India, Indonesia, Papua New Guinea and Sri Lanka to reach the 10,000 people necessary to assess the safety of this new drug combination.

This will be an open label, two-armed study. The two arms are (1) mass drug administration (MDA) with the currently used combination of two-drug regimen (DA) and (2) MDA with triple drug therapy (IDA).

ELIGIBILITY:
In India:

Inclusion Criteria:

1. Age ≥ 5 years, male or female for IDA arm and age > 2 years for DA arm.
2. Able to provide informed consent to participate in the trial (forms to be attached)
3. No evidence of severe or systemic co-morbidities except for features of filarial disease

Exclusion Criteria:

1. Age < 5 years (ivermectin is contraindicated in children below 5 years of age) for IDA arm and age < 2 years for DA arm
2. Pregnant women (DEC, ivermectin and albendazole are contraindicated in pregnancy)
3. Severe chronic illness (for example, chronic renal failure, inability to care for oneself with activities of daily living)
4. History of previous allergy to MDA drugs

For rest of countries:

Inclusion Criteria:

1. Age ≥ 5 years, for IDA and DA arms (males and females).
2. Able to provide informed consent or give parental consent for minors to participate in the trial
3. No evidence of severe or systemic co-morbidities except for features of filarial disease

Exclusion Criteria:

1. Age < 5 years (ivermectin is not approved for use in children less than 5 years of age)
2. Unable to provide informed consent or give parental consent for minors to participate in the trial
3. Pregnant women (DEC, ivermectin and albendazole are not known to be safe for use during pregnancy)
4. Severe chronic illness (chronic renal insufficiency, severe chronic liver disease, or any illness that is severe enough to interfere with activities of daily living)
5. History of previous allergy to MDA drugs

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 23789 (Actual)
Dates: Start 2016-07; Primary Completion 2017-04-27 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by modified CTCAE v4.0 scale | within 7 days of drug administration
  To determine the frequency, type and severity of adverse events following triple-drug therapy Ivermectin, Diethylcarbamazine and Albendazole (IVM+DEC+ALB, IDA) compared to the standard two-drug treatment Diethylcarbamazine and Albendazole (DEC+ALB, DA) in infected and uninfected individuals in a community as assessed by modified CTCAE v4.0 scale.

SECONDARY OUTCOMES:
Number of participants with clearance of microfilaremia (MF) as measured with microfilaremia night blood smear testing (finger prick - 60ul) | baseline (pre-treatment), within 7 days of drug administration and follow up at 12 months
  To compare the efficacy of IDA vs. DA administered in communities for clearance of MF and filarial antigenemia (Ag) in cohort and effectiveness (prevalence) in community settings. A minimum of 21 (70%) of MF-positive participants in each arm will be retested at 12 months post-treatment for antigenemia and microfilaremia. This sample size is adequate to demonstrate superiority of the IDA regimen (assumptions: 90% reduction in MF prevalence after IDA and 60% reduction after DA, 80% power for detecting an effect size of 30%). The primary endpoint for efficacy will be complete clearance of MF 12 months post Mass Drug Administration (MDA). Clearance of filarial antigenemia at 12 months will be a secondary endpoint for the efficacy analysis. Testing of microfilaria is by analyzing 60 microliter (ul) measured volume thick blood smear by finger prick method and results are either positive or negative for MF presence.
Number of participants Filarial Test Strip (FTS) and/or MF positive as tested with FTS and night blood smears with treatment-related adverse events as assessed by modified CTCAE v4.0 scale | baseline (pre-treatment), within 7 days of drug administration and follow up at 12 months
  To assess the presence and intensity of filarial infection on the frequency and severity of adverse events. One year post MDA, all participants who were positive for either microfilaremia or filarial antigenemia during the baseline visit will be tested for filarial antigen using the FTS to assess their response to treatment and to compare the efficacy of the two treatment regimens. Participants with positive FTS will also be tested for nocturnal microfilaremia by blood smear (finger prick - 60ul)
Community acceptance will be measured using on a survey using likert scale questions based on perception of efficacy, intent to participate and relevance of the treatment. | 6-8 months
  Community acceptance will be measured using a survey to community members receiving both the 2-drug and 3-drug treatments during the safety trial. To complement this survey, a series of focus group discussions in the community as well as key informant interviews are proposed with community leaders, health personnel and drug distributors in the same communities to assess perceptions about the 3-drug versus the 2-drug regimen. The community acceptability study will be carried out within one month of the completion of the safety trial. The acceptability score will use a set of likert scale questions based on perception of efficacy, intent to participate and relevance of the treatment. Some of the questions have been inspired by Reimer's Treatment Acceptability Rating form-Revised and general principles of social validity but mostly the questions are not from one particular survey instrument.
Prevalence of STH (hookworm, ascaris, trichuris and strongyloides) as measured by Kato-katz or PCR at baseline and 12 months after treatment | Stool collected at baseline (pre-treatment), 4 weeks (individual response), and 12 months (community prevalence).
  Some sites will include stool sample collections to compare the efficacy of 2 and 3-drug regimens on STH. Stool samples will be analysed using Kato-katz method, as well as PCR.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Weil, MD, Principal Investigator — Washington University School of Medicine; Christopher King, MD PHD, Principal Investigator — Case Western Reserve University
Locations (4):
- Ministere de la Sante Publique et de la Population, Port-au-Prince, Haiti
- Vector Control Research Centre, Puducherry, India
- Universitas Indonesia, Jakarta, Indonesia
- Papua New Guinea Institute for Medical Research, Madang, Papua New Guinea

IPD SHARING:
Plan to Share IPD: Yes
Datasets used for published results will be shared publically through a journal or other open source data repository so that the broader scientific community can access it. Only de-identified data will be shared publicly.
Time Frame: Manuscripts should be submitted for publication no later than one year following the date of the "last patient/last visit". Some DOLF studies include follow-up studies that continue after the primary end point of the study. There is no need to wait for these studies to be completed in order to publish the primary data. (In the case of the IDA studies, safety data should be prepared for publication prior to the acceptability and efficacy studies.)
Access Criteria: Investigators and their supporting institution that conduct research with financial support from Bill & Melinda Gates Foundation (BMGF) will share de-identified data with partner scientists. Results from multiple study sites will be combined so that they can be considered in aggregate. Aggregated data and summary results may be shared with the World Health Org, BMGF, pharmaceutical donors, and others involved in the Global Prog to Eliminate Lymphatic Filariasis even prior to the publication of results. We will follow US National Institutes of Health (NIH) guidelines regarding data sharing with scientists outside of the project. Datasets used for published results will be shared publically through a journal or other open source data repository. De-identified data will be shared outside of DOLF. Data sharing requests from third-parties must have the approval of the local country PI. The study's primary results should be published before data will be shared with third-parties.
URL: http://grants.nih.gov/grants/policy/nihgps/HTML5/section_8/8.2_availability_of_research_results_publications__intellectual_property_rights__and_sharing_research_resources.htm

REFERENCES:
- [Background] World Health Organization (1997). Elimination of lymphatic filariasis as a public health problem - resolution of the executive board of the WHO.
- [Background] Thomsen EK, Sanuku N, Baea M, Satofan S, Maki E, Lombore B, Schmidt MS, Siba PM, Weil GJ, Kazura JW, Fleckenstein LL, King CL. Efficacy, Safety, and Pharmacokinetics of Coadministered Diethylcarbamazine, Albendazole, and Ivermectin for Treatment of Bancroftian Filariasis. Clin Infect Dis. 2016 Feb 1;62(3):334-341. doi: 10.1093/cid/civ882. Epub 2015 Oct 20. PMID 26486704
- [Background] Gyapong JO, Kumaraswami V, Biswas G, Ottesen EA. Treatment strategies underpinning the global programme to eliminate lymphatic filariasis. Expert Opin Pharmacother. 2005 Feb;6(2):179-200. doi: 10.1517/14656566.6.2.179. PMID 15757416
- [Background] 489 Global programme to eliminate lymphatic filariasis: progress report, 2014. Wkly Epidemiol Rec. 2015 Sep 18;90(38):489-504. No abstract available. English, French. PMID 26387149
- [Background] Oscar R, Lemoine JF, Direny AN, Desir L, Beau de Rochars VE, Poirier MJ, Varghese A, Obidegwu I, Lammie PJ, Streit TG, Milord MD. Haiti National Program for the elimination of lymphatic filariasis--a model of success in the face of adversity. PLoS Negl Trop Dis. 2014 Jul 17;8(7):e2915. doi: 10.1371/journal.pntd.0002915. eCollection 2014 Jul. No abstract available. PMID 25032697
- [Background] de Rochars MB, Kanjilal S, Direny AN, Radday J, Lafontant JG, Mathieu E, Rheingans RD, Haddix AC, Streit TG, Beach MJ, Addiss DG, Lammie PJ. The Leogane, Haiti demonstration project: decreased microfilaremia and program costs after three years of mass drug administration. Am J Trop Med Hyg. 2005 Nov;73(5):888-94. PMID 16282299
- [Background] Horton J. Albendazole: a review of anthelmintic efficacy and safety in humans. Parasitology. 2000;121 Suppl:S113-32. doi: 10.1017/s0031182000007290. PMID 11386684
- [Background] Goa KL, McTavish D, Clissold SP. Ivermectin. A review of its antifilarial activity, pharmacokinetic properties and clinical efficacy in onchocerciasis. Drugs. 1991 Oct;42(4):640-58. doi: 10.2165/00003495-199142040-00007. PMID 1723366
- [Background] Edwards G. Ivermectin: does P-glycoprotein play a role in neurotoxicity? Filaria J. 2003 Oct 24;2 Suppl 1(Suppl 1):S8. doi: 10.1186/1475-2883-2-S1-S8. PMID 14975065
- [Background] Ottesen EA, Campbell WC. Ivermectin in human medicine. J Antimicrob Chemother. 1994 Aug;34(2):195-203. doi: 10.1093/jac/34.2.195. PMID 7814280
- [Background] Awadzi K, Edwards G, Duke BO, Opoku NO, Attah SK, Addy ET, Ardrey AE, Quartey BT. The co-administration of ivermectin and albendazole--safety, pharmacokinetics and efficacy against Onchocerca volvulus. Ann Trop Med Parasitol. 2003 Mar;97(2):165-78. doi: 10.1179/000349803235001697. PMID 12803872
- [Background] Ottesen EA. Efficacy of diethylcarbamazine in eradicating infection with lymphatic-dwelling filariae in humans. Rev Infect Dis. 1985 May-Jun;7(3):341-56. doi: 10.1093/clinids/7.3.341. PMID 3895352
- [Background] Noroes J, Dreyer G, Santos A, Mendes VG, Medeiros Z, Addiss D. Assessment of the efficacy of diethylcarbamazine on adult Wuchereria bancrofti in vivo. Trans R Soc Trop Med Hyg. 1997 Jan-Feb;91(1):78-81. doi: 10.1016/s0035-9203(97)90405-3. PMID 9093637
- [Derived] Laman M, Tavul L, Karl S, Kotty B, Kerry Z, Kumai S, Samuel A, Lorry L, Timinao L, Howard SC, Makita L, John L, Bieb S, Wangi J, Albert JM, Payne M, Weil GJ, Tisch DJ, Bjerum CM, Robinson LJ, King CL. Mass drug administration of ivermectin, diethylcarbamazine, plus albendazole compared with diethylcarbamazine plus albendazole for reduction of lymphatic filariasis endemicity in Papua New Guinea: a cluster-randomised trial. Lancet Infect Dis. 2022 Aug;22(8):1200-1209. doi: 10.1016/S1473-3099(22)00026-3. Epub 2022 May 6. PMID 35533701
- [Derived] Tavul L, Laman M, Howard C, Kotty B, Samuel A, Bjerum C, O'Brian K, Kumai S, Amuga M, Lorry L, Kerry Z, Kualawi M, Karl S, Makita L, John LN, Bieb S, Wangi J, Weil GJ, Goss CW, Tisch DJ, Pomat W, King CL, Robinson LJ. Safety and efficacy of mass drug administration with a single-dose triple-drug regimen of albendazole + diethylcarbamazine + ivermectin for lymphatic filariasis in Papua New Guinea: An open-label, cluster-randomised trial. PLoS Negl Trop Dis. 2022 Feb 9;16(2):e0010096. doi: 10.1371/journal.pntd.0010096. eCollection 2022 Feb. PMID 35139070
- [Derived] Supali T, Djuardi Y, Christian M, Iskandar E, Alfian R, Maylasari R, Destani Y, Lomiga A, Minggu D, Lew D, Bogus J, Weil GJ, Fischer PU. An open label, randomized clinical trial to compare the tolerability and efficacy of ivermectin plus diethylcarbamazine and albendazole vs. diethylcarbamazine plus albendazole for treatment of brugian filariasis in Indonesia. PLoS Negl Trop Dis. 2021 Mar 29;15(3):e0009294. doi: 10.1371/journal.pntd.0009294. eCollection 2021 Mar. PMID 33780481
- [Derived] Weil GJ, Bogus J, Christian M, Dubray C, Djuardi Y, Fischer PU, Goss CW, Hardy M, Jambulingam P, King CL, Kuttiat VS, Krishnamoorthy K, Laman M, Lemoine JF, O'Brian KK, Robinson LJ, Samuela J, Schechtman KB, Sircar A, Srividya A, Steer AC, Supali T, Subramanian S; DOLF IDA Safety Study Group. The safety of double- and triple-drug community mass drug administration for lymphatic filariasis: A multicenter, open-label, cluster-randomized study. PLoS Med. 2019 Jun 24;16(6):e1002839. doi: 10.1371/journal.pmed.1002839. eCollection 2019 Jun. PMID 31233507

DOCUMENTS (4):
  • Study Protocol: India specific protocol (2017-09-20): https://cdn.clinicaltrials.gov/large-docs/36/NCT02899936/Prot_000.pdf
  • Study Protocol and Informed Consent Form: Papua New Guinea specific protocol + ICF (2017-07-05): https://cdn.clinicaltrials.gov/large-docs/36/NCT02899936/Prot_ICF_001.pdf
  • Study Protocol and Informed Consent Form: Haiti specific protocol + ICF (2017-07-05): https://cdn.clinicaltrials.gov/large-docs/36/NCT02899936/Prot_ICF_002.pdf
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form: Indonesia specific protocol + ICF (2017-05-24): https://cdn.clinicaltrials.gov/large-docs/36/NCT02899936/Prot_SAP_ICF_003.pdf